CLINICAL TRIAL: NCT03386383
Title: mHealth Physical Activity Intervention for Survivors of Adolescent and Young Adult Cancers
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LCCC1709
Record Dates: First submitted 2017-11-13; First posted 2017-12-29 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Physical Activity
Keywords: adolescent and young adult; cancer survivor
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Masking Description: 4
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive an initial individual session, physical activity tracker, weekly behavioral lessons, tailored feedback summaries, and access to a Facebook group immediately after baseline assessments.
  Interventions: Behavioral: Intervention
- Wait List Control (No Intervention): Participants will receive a physical activity tracker and be advised to maintain their current activity. After 3 months, participants will receive an initial individual session, weekly behavioral lessons, tailored feedback summaries, and access to a Facebook group.

INTERVENTIONS:
Behavioral: Intervention — Individual session, physical activity tracker, online intervention
  Arms: Intervention

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability, and gather preliminary data on outcomes of a 3-month mHealth intervention to promote physical activity among adolescent and young adult (AYA) cancer survivors compared to a delayed intervention control group.

DETAILED DESCRIPTION:
Adolescent and young adult (AYA) survivors are not meeting recommended physical activity guidelines for cancer survivors, and few interventions to date have focused specifically on promoting physical activity among AYAs or capitalized on new technologies to deliver them. This is a pilot randomized controlled trial (RCT) to examine the feasibility, acceptability, and gather preliminary data on outcomes of a 3-month mHealth intervention to promote PA among AYA survivors compared to a delayed intervention control group. This project will focus on how to best integrate self-monitoring with wearable trackers, increase self-efficacy, enhance autonomous motivation, and promote social support in a mobile health behavioral intervention that promotes moderate-to-vigorous intensity physical activity (MVPA) among AYA survivors. Participants will be AYA cancer survivors (N=60), diagnosed at age 15 or older and currently age 18-39. AYA cancer survivors will be recruited from the three comprehensive cancer centers in North Carolina to participate in this study. The behavioral intervention will consist of an activity tracker, Facebook group, weekly email lessons, and weekly tailored feedback emails. Assessments of objectively-measured physical activity and other outcomes will be completed at baseline, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer (excluding basal cell skin cancer) at age 15 or older
* Currently age 18-39
* Are 0 to 10 years post active cancer treatment (i.e., current hormonal treatments or maintenance therapies are permissible)
* Able to speak, read and write English
* Have access to the Internet and computer on at least a weekly basis
* Possession and usage of an Internet e-mail address or willingness to sign up for a free email account
* Have active Facebook account
* Willing to be randomized to either arm

Exclusion Criteria:

* History of heart attack or stroke within past 6 months
* Untreated hypertension, hyperlipidemia, or diabetes, unless permission is provided by their health care provider
* Have a pre-existing medical condition(s) or contraindications that preclude adherence to an unsupervised exercise program, including cardiovascular disease, heart failure, pulmonary conditions, renal disease, and severe orthopedic conditions
* Are already adhering to the American Cancer Society's recommendation of ≥150 minutes of moderate-intensity exercise per week (<150 minutes/week)
* Current participation in another physical activity or weight control program
* Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months
* Plans for major surgery (e.g., breast reconstruction) during the study time frame

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Accrual rate | Through completion of study enrollment, an average of 6 months.
  Number of participants who agreed to participate divided by the number of months of recruitment.
Participation rate | Through completion of study enrollment, an average of 6 months.
  Percentage of eligible participants who agreed to participate.
Retention rate at 3 months | 3 months
  Number of intervention participants who completed 3-month measures divided by the number who consented to participate.

SECONDARY OUTCOMES:
Retention rate at 6 months | 6 months
  Number of intervention participants who completed 6-month measures divided by the number randomized to the intervention group.
Satisfaction with intervention | 6 months
  Ratings of satisfaction with the intervention, as measured by satisfaction questionnaire.
Adherence to physical activity monitoring | Through study completion, 6 months
  Number of days physical activity tracked, as measured by Fitbit.
Physical activity: objective | Baseline, 3 months, 6 months
  Change in objective levels of physical activity, as measured by accelerometry (Actigraph), from baseline to 3 months, and 3 months to 6 months.
Physical activity: self-report | Baseline, 3 months, 6 months
  Change in self-report levels of physical activity, as measured by the Godin Leisure Time Exercise Questionnaire, from baseline to 3 months, and 3 months to 6 months.
Sedentary behavior: self-report | Baseline, 3 months, 6 months
  Change in self-report levels of sedentary behavior, as measured by the Marshall Sitting Time Questionnaire, from baseline to 3 months, and 3 months to 6 months.
Weight | Baseline, 3 months, 6 months
  Change in self-reported weight, from baseline to 3 months, and 3 months to 6 months.
Intrinsic motivation | Baseline, 3 months, 6 months
  Change in intrinsic motivation, as measured by the intrinsic motivation subscale of the Treatment Self-Regulation Questionnaire for Exercise, from baseline to 3 months, and 3 months to 6 months. Responses to four items comprising intrinsic motivation subscale are averaged to yield a score from 1 to 7, with higher values representing higher intrinsic motivation.
Self-efficacy for exercise | Baseline, 3 months, 6 months
  Change in self-efficacy for exercise, as measured by the Self-Efficacy and Exercise Habits Survey, from baseline to 3 months, and 3 months to 6 months. Responses for two subscales (Sticking to it, Making time for exercise) are averaged to yield a score from 1 to 5, with higher values representing higher self-efficacy for exercise.
Social support for exercise | Baseline, 3 months, 6 months
  Change in social support for exercise, as measured by the Social Support for Exercise Survey, from baseline to 3 months, and 3 months to 6 months. Responses for three factors (Family participation, Friend participation, Friends on social networking sites participation), ranging from 1 to 5, are summed, with higher values representing higher social support for exercise.

OTHER OUTCOMES:
Posttraumatic growth | Baseline, 3 months, 6 months
  Change in posttraumatic growth, as measured by the Short Form of the Posttraumatic Growth Inventory, from baseline to 3 months, and 3 months to 6 months. Responses range from 0 to 5 and yield an overall score and subscale scores for relating to others, new possibilities, personal strength, spiritual change, and appreciation of life. Items are summed, with higher scores reflecting more positive change (i.e., posttraumatic growth).
Positive psychosocial illness impact | Baseline, 3 months, 6 months
  Changes in positive psychosocial impact of illness, as measured by the PROMIS Psychosocial Illness Impact - Positive (4a), from baseline to 3 months, and 3 months to 6 months. Responses to the 4-item short from range from 1 to 5. Items are summed, with higher scores reflecting more positive psychosocial impact.
Negative psychosocial illness impact | Baseline, 3 months, 6 months
  Changes in positive psychosocial impact of illness, as measured by the PROMIS Psychosocial Illness Impact - Negative (4a), from baseline to 3 months, and 3 months to 6 months. Responses to the 4-item short from range from 1 to 5. Items are summed, with higher scores reflecting more negative psychosocial impact.
Positive affect | Baseline, 3 months, 6 months
  Changes in positive affect, as measured by the NIH Toolbox Positive Affect Short Form, from baseline to 3 months, and 3 months to 6 months.
Social network orientation | Baseline, 3 months, 6 months
  Changes in positive affect, as measured by the Network Orientation Scale, from baseline to 3 months, and 3 months to 6 months. Responses to 20 items range from 1 to 4. Items are summed (range: 20 to 80), with higher scores representing a more negative social network orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Carmina G. Valle, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; John M. Salsman, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No